CLINICAL TRIAL: NCT02805582
Title: Area of Sensory Loss, Onset Time and Duration of Two Different Ultrasound Guided Intercostobrachial Nerve Blocks for Vascular Access Surgery of the Upper Arm
Brief Title: Ultrasound Guided Intercostobrachial Nerve Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Christoph Ilies (Other)
Responsible Party: Sponsor-Investigator, Dr. Christoph Ilies, Dr. med., Marienhospital Stuttgart
Organization: Marienhospital Stuttgart (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: iCobra 2016
Record Dates: First submitted 2016-04-28; First posted 2016-06-20 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Anaesthesia
Keywords: Peripheral Nerve Block

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anterior musculus serratus block (Active Comparator): Proximal nerve block above the second intercostal space between Musculus serratus anterior and Musculus pectoralis minor.
  Intervention: 10ml ropivacain 0.5%
  Interventions: Drug: 10ml ropivacain 0.5%
- Subpectoral block (Active Comparator): Distal nerve block under the Musculus pectoralis major at the medial border of the axillary triangle.
  Intervention: 10ml ropivacain 0.5%
  Interventions: Drug: 10ml ropivacain 0.5%

INTERVENTIONS:
Drug: 10ml ropivacain 0.5% — Ultrasound guided nerve block
  Other Names: ropivacain Sintetica 0.5%

SUMMARY:
The intercostobrachial nerve underlies many anatomical variations. For surgery of the upper arm the axilla is usually not anaesthetized by a brachial plexus block, which therefore needs to be completed by an intercostobrachial nerve block. The optimal access for an ultrasound guided block of the intercostobrachial nerve is not yet known. The investigators compare a proximal and a more distal approach to the nerve referred to onset time, sensory blocked area and duration.

DETAILED DESCRIPTION:
The participants will be randomized into two groups:

Group one receives a modified PECS 2 (thoracic wall) block above the second intercostal space with injection between the Musculus serratus anterior and Musculus pectoralis minor.

Group 2 receives a subpectoral block under the pectoralis major muscle at the medial boarder of the axillary triangle.

ELIGIBILITY:
Inclusion Criteria:

* patients planned for vascular access surgery of the upper arm
* surgery planned under regional anaesthesia

Exclusion Criteria:

* patients refusal
* age under 18
* allergy against local anaesthetics
* polyneuropathies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Blocked area in squared cm | Assessment 30 minutes after intervention
  Area of sensory loss to pin prick test

SECONDARY OUTCOMES:
Block onset time in minutes | Complete timeframe of 45 minutes with testing every 5 minutes
  Onset time of complete analgesia. Assessment by pin prick test in the middle of the axilla
Block duration in minutes | Assessment every 30 minutes for 8 hours after nerve block
  Complete analgesia to pin prick in the middle of the axilla
The pain numeric rating scale (NRS) during surgical manipulation in the axilla | From beginning to end of surgery. Estimated mean duration of 90 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Marienhospital Stuttgart, Dpt. of Anaesthesiology, Stuttgart, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No